CLINICAL TRIAL: NCT00645827
Title: Use of an Insulin Infusion Conversion Equation (IICE) to Improve Inpatient Glycemic Control: A Randomized Controlled Trial
Brief Title: Use of an Insulin Infusion Conversion Equation (IICE) to Control Blood Glucose in Hospitalized Patients
Acronym: IICE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Responsible Party: Principal Investigator, G. Randy Smith, Jr., M.D., Principal Investigator, Emory University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB00006564
Record Dates: First submitted 2008-03-25; First posted 2008-03-28 (Estimated); Results first posted 2014-09-15 (Estimated); Last update posted 2014-09-15 (Estimated); Status verified 2014-09

CONDITIONS: Glucose, Blood
Keywords: Insulin; Blood Glucose
MeSH Terms: conditions — Insulin Resistance

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Insulin infusion conversion equation (Experimental): Insulin infusion conversion equation is used to determine subcutaneous insulin dosing for first 24 hours after cessation of an IV insulin infusion.
  Interventions: Other: IICE Dosing
- Control (Active Comparator): Judgment of patient's healthcare provider is used to determine subcutaneous insulin dosing for first 24 hours after cessation of IV insulin infusion.
  Interventions: Other: Healthcare Provider dosing

INTERVENTIONS:
Other: IICE Dosing — Subcutaneous insulin was dosed according to an equation (too long for publication here) which gives the patient's 24 hour SC insulin requirement. If patient was eating, 65% of equation result was given as insulin glargine SC qHS and 35% of equation result was divided evenly between three qAC doses of insulin aspart. If patient was not eating, 100% of ISC was given as insulin glargine. If IV insulin was stopped between 7 AM and 3 PM, 1/2 to 1/3 of scheduled insulin glargine dose was given as a one time insulin NPH SC dose at time of IV insulin cessation. Correctional insulin was given as follows: For BG ≥ 150 mg/dL, (BG-100)/X units insulin aspart SC, X = 1500 / (scheduled glargine dose + [3 x scheduled aspart dose]). For BG < 70 mg/dL, ½ ampule D50W IV x1 was given.
  Arms: Insulin infusion conversion equation
Other: Healthcare Provider dosing — Twenty-four hour subcutaneous insulin dosing requirement was determined according to the judgment of the patient's healthcare provider. If patient was eating, insulin glargine SC qHS and three qAC doses of insulin aspart was given according to the judgment of the patients's healthcare provider. If patient was not eating, 100% of insulin was given as insulin glargine. If IV insulin was stopped between 7 AM and 3 PM, 1/2 to 1/3 of scheduled insulin glargine dose was given as a one time insulin NPH SC dose at time of IV insulin cessation. Correctional insulin was given as follows: For BG ≥ 150 mg/dL, (BG-100)/X units insulin aspart SC, X = 1500 / (scheduled glargine dose + [3 x scheduled aspart dose]). For BG < 70 mg/dL, ½ ampule D50W IV x1 was given.
  Arms: Control

SUMMARY:
Insulin infusions are commonly used in hospitalized diabetics to control blood sugar, and they are effective. However, insulin infusions require the use of limited resources. Insulin infusions are therefore changed to insulin shots as a patient recovers. Once an insulin infusion is stopped and shots are started, blood sugar control is harder to maintain. This is, in part, because physicians have different ideas on how to dose insulin shots in hospitalized patients. A math equation has been developed by the research staff that attempts to predict the effective doses of insulin shots in patients whose insulin infusion have just been stopped. The math equation was developed for patients with type 2 diabetes mellitus. In this study, all patients will be treated with the same type of insulin shots, with doses of the insulin shots chosen either by the math equation or by the judgment of the patient's physician. The study will then follow blood sugar values for 24 hours to see if the math equation is effective. If the equation is proven to be effective, a new tool will exist for physicians to determine the best dose of insulin shots for type 2 diabetics. Such a tool would, in turn, allow for widespread use of insulin infusions to determine a patient's insulin needs before discharge from the hospital. Blood sugar control for type 2 diabetics that are inpatient or outpatient would improve as a result, with potentially far reaching public health benefits.

ELIGIBILITY:
Inclusion Criteria:

* Inpatients at an urban, mixed academic and community tertiary care hospital who were on IV insulin were enrolled.
* Patients were taken from medical, general surgical, and cardiothoracic services, and were located both inside and outside the intensive care unit (ICU).

Exclusion Criteria:

* At time of enrollment, patients with type I diabetes mellitus,
* active acute or chronic pancreatitis,
* history of pancreatic surgery,
* use of a self-titratable insulin pump, or
* history of β-islet cell transplantation were excluded.
* At time of randomization, patients with insulin drip rates ≤ 2 units/hr, ∆ in serum creatinine of > 20% in previous 24 hours, or
* those without caloric intake while on IV insulin were excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2008-01; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gregory R Smith, Jr., MD, Principal Investigator — Emory University
Locations (1):
- Emory Crawford Long Hospital, Atlanta, Georgia, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were enrolled between April 2008 to February 2009.
Pre-assignment Details: 78 subjects consented. 3 subjects excluded at screening. Of the 75 subjects remaining, only 57 subjects seen by the principal investigator (PI) because the patient's healthcare provider had to call the PI right before the intravenous insulin infusion (III) was discontinued. PI excluded 26 more subjects at III cessation--31 subjects randomized.
Period: Overall Study
Arm/Group | Insulin Infusion Conversion Equation | Control
Started | 14 | 17
Completed | 14 | 17
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Insulin Infusion Conversion Equation | Control | Total
Number analyzed (Participants) | 14 | 17 | 31
Age, Customized [Number; unit: participants] — Age > 18 years old
  participants
    Age > 18 years old | 14 | 17 | 31
Sex/Gender, Customized [Number; unit: participants] — Gender not collected
  participants
    Unknown | 14 | 17 | 31
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 9 | 10 | 19
  White | 5 | 7 | 12
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 14 | 17 | 31

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Blood Glucose Values Within 80-140 mg/dL
Description: Fingerstick glucose measurements were obtained up to six times for each participant. Percentage of blood glucose values within the target range of 80-140 mg/dL
Time Frame: Within 24 hours after cessation of IV insulin
Measure: Number; unit: percentage of blood glucose values
Arm/Group | Insulin Infusion Conversion Equation | Control
Number analyzed (Participants) | 14 | 17
percentage of blood glucose values | 54.8 [0.42 to 0.68] | 21.2 [0.1 to 0.33]

2. Secondary Outcome: Hypoglycemia (Serum Blood Glucose < 70 mg/dL)
Time Frame: Within 24 hours after cessation of IV insulin
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | Insulin Infusion Conversion Equation | Control
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/17
Other Adverse Events (participants affected / at risk) | 0/14 | 0/17

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes